CLINICAL TRIAL: NCT02035137
Title: NANT 2011- 01: Randomized Phase II Pick the Winner Study of 131I-MIBG, 131I-MIBG With Vincristine and Irinotecan, or 131I-MIBG With Vorinostat for Resistant/Relapsed Neuroblastoma
Brief Title: 131I-MIBG Alone VS. 131I-MIBG With Vincristine and Irinotecan VS131I-MIBG With Vorinostat
Acronym: N2011-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N2011-01
Record Dates: First submitted 2014-01-07; First posted 2014-01-14 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — 3-Iodobenzylguanidine; Vincristine; Irinotecan; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Single-Agent 131I-MIBG (Active Comparator): Single-agent 131I-MIBG (Arm A) 18 mCi/kg 131I-MIBG on Day 1 and autologous stem cell infusion on Day 15.
  Interventions: Radiation: 131I-MIBG
- 131I-MIBG with Vincristine/Irinotecan (Active Comparator): Vincristine / irinotecan / 131I-MIBG (Arm B): vincristine 2 mg/m2 (maximum dose 2 mg) intravenously on Day 0; irinotecan 50 mg/m2 (maximum dose 100 mg) intravenously on Days 0 to 4. Patients will also receive diarrhea prophylaxis with cefixime 8 mg/kg/day orally on Days -1 to +6. 131I-MIBG, 18 mCi/kg on Day 1 and autologous stem cell infusion on Day 15.
  Interventions: Radiation: 131I-MIBG; Drug: Vincristine; Drug: Irinotecan
- 131I-MIBG with Vorinostat (Active Comparator): Vorinostat / 131I-MIBG (Arm C); vorinostat 180 mg/m2 (maximum dose 400 mg) orally once daily on Days -1 to +12 (14 total doses). 131I-MIBG, 18 mCi/kg on Day 1 and autologous stem cell infusion on Day 15.
  Interventions: Radiation: 131I-MIBG; Drug: Vorinostat

INTERVENTIONS:
Radiation: 131I-MIBG
  Other Names: 131I-Metaiodobenzylguanidine; Iobenguane sulfate; m-Iodobenzylguanidine sulfate; MIBG
Drug: Vincristine
  Arms: 131I-MIBG with Vincristine/Irinotecan
Drug: Irinotecan
  Arms: 131I-MIBG with Vincristine/Irinotecan
Drug: Vorinostat
  Other Names: Zolinza
  Arms: 131I-MIBG with Vorinostat

SUMMARY:
This study will compare three treatment regimens containing metaiodobenzylguanidine (MIBG) and compare their effects on tumor response and associated side effects, to determine if one therapy is better than the other for people diagnosed with relapsed or persistent neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 24 months and < 30 years of age when registered on study.
* Patients must have relapsed neuroblastoma, refractory neuroblastoma that had less than a partial response to standard treatment or persistent neuroblastoma that had at least a partial response to frontline therapy frontline therapy with > 3 residual lesions on end-induction MIBG scan.
* Patients must have evidence of MIBG uptake into tumor at ≥ one site within 4 weeks prior to entry on study and subsequent to any intervening therapy.
* Patients must have adequate heart, kidney, liver and bone marrow function. Patients who have bone marrow disease must still have adequate bone marrow function to enter the study.
* Patients must have a dose of unpurged peripheral blood stem cells is 2.0 x 106 viable CD34+ cells/kg available.

Exclusion Criteria:

* They have had previous I-131 MIBG therapy
* They have other medical problems that could get much worse with this treatment.
* They are pregnant or breast feeding.
* They have a history of a venous or arterial thrombosis that was not associated to a central line.
* They have active infections such as hepatitis or fungal infections.
* They have active diarrhea.
* They have had an allogeneic stem cell transplant (received stem cell from someone else)
* They can't cooperate with the special precautions that are needed for this trial.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2014-07; Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven DuBois, MD, Study Chair — Dana-Farber Cancer Institute
Locations (14):
- United States (13):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile Salter Packer Children's Hospital, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children Hospital of Colorado, Aurora, Colorado
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - University of Chicago, Comer Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - C.S Mott Children's Hospital, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Healthcare System, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] DuBois SG, Granger MM, Groshen S, Tsao-Wei D, Ji L, Shamirian A, Czarnecki S, Goodarzian F, Berkovich R, Shimada H, Villablanca JG, Vo KT, Pinto N, Mosse YP, Maris JM, Shusterman S, Cohn SL, Goldsmith KC, Weiss B, Yanik GA, Twist CJ, Irwin MS, Haas-Kogan DA, Park JR, Marachelian A, Matthay KK. Randomized Phase II Trial of MIBG Versus MIBG, Vincristine, and Irinotecan Versus MIBG and Vorinostat for Patients With Relapsed or Refractory Neuroblastoma: A Report From NANT Consortium. J Clin Oncol. 2021 Nov 1;39(31):3506-3514. doi: 10.1200/JCO.21.00703. Epub 2021 Jul 16. PMID 34270348

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-Agent 131I-MIBG: Single-agent 131I-MIBG (Arm A) 18 mCi/kg 131I-MIBG on Day 1 and autologous stem cell infusion on Day 15.
  131I-MIBG
- 131I-MIBG With Vincristine/Irinotecan: Vincristine / irinotecan / 131I-MIBG (Arm B): vincristine 2 mg/m2 (maximum dose 2 mg) intravenously on Day 0; irinotecan 50 mg/m2 (maximum dose 100 mg) intravenously on Days 0 to 4. Patients will also receive diarrhea prophylaxis with cefixime 8 mg/kg/day orally on Days -1 to +6. 31I-MIBG, 18 mCi/kg on Day 1 and autologous stem cell infusion on Day 15.
  131I-MIBG
  Vincristine
  Irinotecan
- 131I-MIBG With Vorinostat: Vorinostat / 131I-MIBG (Arm C); vorinostat 180 mg/m2 (maximum dose 400 mg) orally once daily on Days -1 to +12 (14 total doses). 131I-MIBG, 18 mCi/kg on Day 1 and autologous stem cell infusion on Day 15.
  131I-MIBG
  Vorinostat
Period: Overall Study
Arm/Group | Single-Agent 131I-MIBG | 131I-MIBG With Vincristine/Irinotecan | 131I-MIBG With Vorinostat
Started | 38 | 37 | 39
Completed | 36 | 35 | 34
Not Completed | 2 | 2 | 5
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Ineligible | 0 | 1 | 2
Not completed — Disease progression prior to treatment start | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 111 patients described as baseline participants removes the 3 ineligible patients as provided in the initial row of the participant flow module.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-Agent 131I-MIBG | 131I-MIBG With Vincristine/Irinotecan | 131I-MIBG With Vorinostat | Total
Number analyzed (Participants) | 38 | 36 | 37 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 34 | 36 | 107
  Between 18 and 65 years | 1 | 2 | 1 | 4
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 16 | 52
  Male | 19 | 19 | 21 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 10 | 24
  Not Hispanic or Latino | 30 | 27 | 25 | 82
  Unknown or Not Reported | 1 | 2 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 3 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 4 | 4 | 4 | 12
  White | 26 | 23 | 23 | 72
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 4 | 5 | 7 | 16
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 1 | 3
  United States | 37 | 35 | 36 | 108

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response After One Course of Therapy
Description: To identify the MIBG treatment regimen associated with the highest overall response rate after one course of treatment on the three arms. The response evaluation was based on central review (intent to treat analysis). Responders defined as meeting CR/MRD/PR criteria. Response was based on NANT response criteria v1.2 (https://doi.org/10.1002/pbc.26940). RECST 1.1 criteria was used for measurable tumors with PR criteria > 30% decrease in target tumor size. Curie score was used with PR criteria > 50% decrease in Curie score. Complete Response- disappearance of all target lesions, Curie score of 0 and no detectable bone marrow disease. Overall Response (OR)=CR+PR.
Time Frame: 43-50 days from study day 1
Population: Number of eligible randomized patients who received 131-I-MIBG therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Agent 131I-MIBG | 131I-MIBG With Vincristine/Irinotecan | 131I-MIBG With Vorinostat
Number analyzed (Participants) | 36 | 35 | 34
Participants | 5 | 5 | 11

2. Secondary Outcome: Number of Participants With Grade 3 or Greater Non-hematologic Toxicities
Description: Compare toxicity profiles for grade 3 or greater toxicities associated with each of 131I-MIBG treatment regimens; single-agent 131I-MIBG; Vincristine/Irinotecan/131I-MIBG; or Vorinostat/131I-MIBG
Time Frame: All toxicities from enrollment through 30 days following end of protocol therapy, an average of 6 months
Population: Patients who were eligible, randomized, and received 131I-MIBG treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single-Agent 131I-MIBG | 131I-MIBG With Vincristine/Irinotecan | 131I-MIBG With Vorinostat
Number analyzed (Participants) | 36 | 35 | 34
Participants | 7 | 17 | 12

ADVERSE EVENTS:
Time Frame: All adverse events from enrollment through 30 days following end of protocol therapy, an average of 6 months
Description: The 111 patients described as participants do not include the 3 ineligible patients as provided in the initial row of the participant flow module
Arm/Group | Single-Agent 131I-MIBG | 131I-MIBG With Vincristine/Irinotecan | 131I-MIBG With Vorinostat
All-Cause Mortality (participants affected / at risk) | 11/38 | 17/36 | 18/37
Serious Adverse Events (participants affected / at risk) | 6/38 | 12/36 | 5/37
Other Adverse Events (participants affected / at risk) | 37/38 | 35/36 | 35/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Agent 131I-MIBG (N=38) | 131I-MIBG With Vincristine/Irinotecan (N=36) | 131I-MIBG With Vorinostat (N=37)
10000060-Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
10000081-Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0
10002272-Anemia (Blood and lymphatic system disorders) | 4 | 6 | 0
10002646-Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 0
10003988-Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
10007810-Catheter related infection (Infections and infestations) | 1 | 1 | 0
10010774-Constipation (Gastrointestinal disorders) | 0 | 2 | 0
10011224-Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
10012174-Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0
10012727-Diarrhea (Gastrointestinal disorders) | 0 | 3 | 0
10013781-Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
10016256-Fatigue (General disorders) | 0 | 3 | 1
10016288-Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 0
10016558-Fever (General disorders) | 1 | 1 | 2
10019211-Headache (Nervous system disorders) | 0 | 1 | 0
10020943-Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 1
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
10021018-Hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 1
10021038-Hyponatremia (Metabolism and nutrition disorders) | 0 | 4 | 0
10021059-Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 1
10021143-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
10021328-Ileus (Gastrointestinal disorders) | 0 | 1 | 0
10022437-Insomnia (Psychiatric disorders) | 0 | 1 | 0
10024264-Lethargy (Nervous system disorders) | 0 | 2 | 0
10025256-Lymphocyte count decreased (Investigations) | 1 | 3 | 0
10028411-Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
10028813-Nausea (Gastrointestinal disorders) | 0 | 2 | 0
10029366-Neutrophil count decreased (Investigations) | 0 | 4 | 0
10033425-Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
10034960-Photophobia (Eye disorders) | 0 | 1 | 0
10035528-Platelet count decreased (Investigations) | 2 | 5 | 1
10035598-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
10040752-Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
10047700-Vomiting (Gastrointestinal disorders) | 0 | 4 | 1
10047900-Weight loss (Investigations) | 0 | 3 | 0
10048677-Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
10049182-White blood cell decreased (Investigations) | 1 | 5 | 1
10049737-Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
10059827-Rhinitis infective (Infections and infestations) | 1 | 0 | 0
CLOSTRIDIUM DIFFICILE (Infections and infestations) | 0 | 1 | 0
ENTEROBACTER CLOCACAE (Infections and infestations) | 0 | 0 | 1
PILONIDAL CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Agent 131I-MIBG (N=38) | 131I-MIBG With Vincristine/Irinotecan (N=36) | 131I-MIBG With Vorinostat (N=37)
10000060-Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 2
10000081-Abdominal pain (Gastrointestinal disorders) | 7 | 11 | 2
10000636-Activated partial thromboplastin time prolonged (Investigations) | 3 | 2 | 16
10001497-Agitation (Psychiatric disorders) | 0 | 1 | 2
10001551-Alanine aminotransferase increased (Investigations) | 21 | 22 | 17
10001675-Alkaline phosphatase increased (Investigations) | 7 | 2 | 5
10001718-Allergic reaction (Immune system disorders) | 0 | 1 | 0
10001723-Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
10001760-Alopecia (Skin and subcutaneous tissue disorders) | 0 | 5 | 2
10002167-Anal pain (Gastrointestinal disorders) | 1 | 0 | 0
10002272-Anemia (Blood and lymphatic system disorders) | 34 | 33 | 32
10002646-Anorexia (Metabolism and nutrition disorders) | 10 | 15 | 14
10002855-Anxiety (Psychiatric disorders) | 2 | 2 | 3
10003481-Aspartate aminotransferase increased (Investigations) | 23 | 21 | 21
10003988-Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
10005364-Blood bilirubin increased (Investigations) | 3 | 3 | 3
10005886-Blurred vision (Eye disorders) | 1 | 2 | 0
10006002-Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0
10006504-Bruising (Injury, poisoning and procedural complications) | 3 | 1 | 4
10007810-Catheter related infection (Infections and infestations) | 2 | 2 | 1
10007839-CD4 lymphocytes decreased (Investigations) | 1 | 2 | 0
10008496-Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
10008531-Chills (General disorders) | 0 | 1 | 1
10009887-Colitis (Gastrointestinal disorders) | 0 | 0 | 1
10010774-Constipation (Gastrointestinal disorders) | 7 | 11 | 7
10011224-Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 8 | 11
10011368-Creatinine increased (Investigations) | 1 | 1 | 4
10012174-Dehydration (Metabolism and nutrition disorders) | 0 | 7 | 2
10012378-Depression (Psychiatric disorders) | 0 | 1 | 0
10012727-Diarrhea (Gastrointestinal disorders) | 4 | 24 | 8
10013573-Dizziness (Nervous system disorders) | 1 | 2 | 1
10013781-Dry mouth (Gastrointestinal disorders) | 2 | 2 | 3
10013786-Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
10013911-Dysgeusia (Nervous system disorders) | 0 | 0 | 1
10013946-Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
10013963-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
10014020-Ear pain (Ear and labyrinth disorders) | 1 | 2 | 0
10014222-Edema face (General disorders) | 2 | 7 | 2
10014383-Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 3
10015090-Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
10015958-Eye pain (Eye disorders) | 1 | 0 | 0
10016059-Facial pain (General disorders) | 0 | 1 | 1
10016256-Fatigue (General disorders) | 11 | 16 | 12
10016288-Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 0
10016558-Fever (General disorders) | 10 | 10 | 10
10016778-Floaters (Eye disorders) | 1 | 0 | 0
10016791-Flu like symptoms (General disorders) | 1 | 0 | 1
10016825-Flushing (Vascular disorders) | 0 | 0 | 1
10017076-Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
10017577-Gait disturbance (General disorders) | 0 | 0 | 1
10019211-Headache (Nervous system disorders) | 7 | 6 | 5
10019245-Hearing impaired (Ear and labyrinth disorders) | 0 | 2 | 1
10019450-Hematuria (Renal and urinary disorders) | 2 | 2 | 1
10020039-Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
10020587-Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1 | 1
10020639-Hyperglycemia (Metabolism and nutrition disorders) | 7 | 5 | 10
10020647-Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2 | 2
10020670-Hypermagnesemia (Metabolism and nutrition disorders) | 6 | 2 | 7
10020680-Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 2
10020772-Hypertension (Vascular disorders) | 3 | 4 | 3
10020870-Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 4 | 0
10020943-Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 11 | 11
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 8 | 9 | 8
10021005-Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2 | 2
10021018-Hypokalemia (Metabolism and nutrition disorders) | 8 | 10 | 10
10021028-Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 13 | 4
10021038-Hyponatremia (Metabolism and nutrition disorders) | 14 | 15 | 13
10021059-Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 6 | 8
10021097-Hypotension (Vascular disorders) | 1 | 2 | 4
10021114-Hypothyroidism (Endocrine disorders) | 1 | 3 | 1
10021143-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
10021328-Ileus (Gastrointestinal disorders) | 0 | 1 | 0
10022402-INR increased (Investigations) | 2 | 1 | 6
10022437-Insomnia (Psychiatric disorders) | 1 | 2 | 0
10022998-Irritability (General disorders) | 1 | 1 | 0
10024264-Lethargy (Nervous system disorders) | 1 | 4 | 0
10025256-Lymphocyte count decreased (Investigations) | 27 | 28 | 28
10025258-Lymphocyte count increased (Investigations) | 0 | 0 | 1
10025482-Malaise (General disorders) | 2 | 2 | 2
10028130-Mucositis oral (Gastrointestinal disorders) | 1 | 4 | 2
10028411-Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
10028735-Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 6
10028813-Nausea (Gastrointestinal disorders) | 14 | 23 | 13
10028836-Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
10029366-Neutrophil count decreased (Investigations) | 34 | 31 | 31
10030980-Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
10031009-Oral pain (Gastrointestinal disorders) | 2 | 3 | 1
10033371-Pain (General disorders) | 2 | 8 | 4
10033425-Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 6 | 2
10033987-Paresthesia (Nervous system disorders) | 0 | 0 | 1
10034310-Penile pain (Reproductive system and breast disorders) | 2 | 2 | 2
10034620-Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
10034960-Photophobia (Eye disorders) | 2 | 1 | 0
10035528-Platelet count decreased (Investigations) | 35 | 34 | 34
10035598-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
10036790-Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
10037032-Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
10037087-Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
10037868-Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
10038064-Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
10038072-Rectal pain (Gastrointestinal disorders) | 0 | 1 | 0
10038695-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
10040047-Sepsis (Infections and infestations) | 0 | 0 | 1
10040741-Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
10040752-Sinus tachycardia (Cardiac disorders) | 4 | 7 | 5
10040865-Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
10040872-Skin infection (Infections and infestations) | 1 | 0 | 0
10041232-Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
10041349-Somnolence (Nervous system disorders) | 0 | 0 | 1
10041367-Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 2
10042112-Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0
10042458-Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
10044055-Toothache (Gastrointestinal disorders) | 1 | 0 | 0
10045158-Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
10046300-Upper respiratory infection (Infections and infestations) | 1 | 4 | 1
10046539-Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0
10046555-Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
10046571-Urinary tract infection (Infections and infestations) | 3 | 0 | 0
10047700-Vomiting (Gastrointestinal disorders) | 15 | 21 | 20
10047900-Weight loss (Investigations) | 1 | 9 | 5
10048677-Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
10048994-Bladder spasm (Renal and urinary disorders) | 1 | 2 | 0
10049182-White blood cell decreased (Investigations) | 32 | 33 | 30
10050068-Edema limbs (General disorders) | 1 | 0 | 1
10051792-Infusion related reaction (General disorders) | 1 | 0 | 1
10054482-Neck edema (General disorders) | 0 | 1 | 1
10056910-GGT increased (Investigations) | 1 | 1 | 2
10061322-Optic nerve disorder (Eye disorders) | 0 | 0 | 1
10062225-Urinary tract pain (Renal and urinary disorders) | 2 | 0 | 0
10062466-Localized edema (General disorders) | 1 | 0 | 0
10062501-Non-cardiac chest pain (General disorders) | 0 | 0 | 1
10062572-Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
10065764-Mucosal infection (Infections and infestations) | 0 | 1 | 1
10065776-Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
10065780-Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
10065838-Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0
10065973-Iron overload (Metabolism and nutrition disorders) | 1 | 0 | 0
10066874-Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
ADJUSTMENT DISORDER (Psychiatric disorders) | 1 | 0 | 0
C DIFFICILE (Infections and infestations) | 0 | 1 | 0
CATHETER RELATED PAIN (Renal and urinary disorders) | 0 | 1 | 0
CHEST DISCOMFORT, ""TIGHTNESS"" (General disorders) | 0 | 1 | 0
CLOSTRIDIUM DIFICILE (Infections and infestations) | 0 | 1 | 0
CONCERN FOR DISEASE PROGRESSION AS INDICATED BY INTERVAL INCREASE IN THE SIZE OF HER OCCIPITAL MASS (General disorders) | 1 | 0 | 0
DISEASE PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
DRY CRACKED LIPS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
ENTEROBACTER CLOACAE (Infections and infestations) | 1 | 0 | 0
HYPERPHOSPHATEMIA (Investigations) | 1 | 0 | 1
INFLUENZA A (Infections and infestations) | 0 | 0 | 1
INJECTED EYE (Eye disorders) | 0 | 1 | 0
INJURY TO LEFT WRIST (Injury, poisoning and procedural complications) | 1 | 0 | 0
IRRITATION AROUND CATHETER (General disorders) | 0 | 1 | 0
JAW PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
KETONURIA (Renal and urinary disorders) | 0 | 1 | 0
MALNUTRITION - ANOREXIA (Metabolism and nutrition disorders) | 0 | 1 | 0
MULTIPLE BACTERIAL INFECTIONS (ENTEROBACTER, CITROBACTER, KLEBSIELLA, GPC, GVC) (Infections and infestations) | 0 | 0 | 1
MURMUR (Cardiac disorders) | 0 | 0 | 1
ODD/ANXIETY (Psychiatric disorders) | 0 | 1 | 0
PAIN (General disorders) | 0 | 1 | 0
PAIN IN EXTREMITY -RIGHT FOOT (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
PAIN RIGHT SIDE JAW (General disorders) | 0 | 1 | 0
PAIN, LEG (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
PAPULOERYTHEMATOUS LESIONS - LEFT CHEEK (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PARAPHIMOSIS (Reproductive system and breast disorders) | 1 | 0 | 0
PAROTIDITIS (Infections and infestations) | 1 | 0 | 0
PILONIDAL CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
RASH - CHEST (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
RASH - UPPER CHEST AND BACK (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
RESPIRATORY DEPRESSION FROM SEDATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RHINOVIRUS (Infections and infestations) | 1 | 0 | 0
RIB PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SCRATCH (Injury, poisoning and procedural complications) | 0 | 1 | 0
STOMACH CRAMPING (Gastrointestinal disorders) | 0 | 1 | 0
UNCOMPENSATED HYPOTHYROIDISM (Endocrine disorders) | 0 | 1 | 0
URETHRAL TRAUMA (Renal and urinary disorders) | 0 | 0 | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT02035137/Prot_SAP_ICF_000.pdf